CLINICAL TRIAL: NCT04119973
Title: A Multicenter Prospective Study of Application of Platelet Mapping in Acute-on-chronic-liver Failure in China
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southwest Hospital, China (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Xiangya Hospital of Central South University (Other); Taihe Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 009
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-05

CONDITIONS: Thrombelastography; Acute on Chronic Liver Failure; Platelet; Multicenter Prospective Study
Keywords: Thrombelastography; Acute on Chronic Liver Failure; Platelet; Multicenter Prospective Study
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard treatment — standard medical treatment

SUMMARY:
Ineffective hemostasis or a paradoxical prothrombotic state of Acute-on-chronic liver disease (ACLF) has been well established. Thrombelastography measures the dynamics of thrombin production and provides a global assessment of coagulation incorporating the cumulative effect of the interactions at various levels between plasma components and cellular component of coagulation. And through the platelet mapping, it can help provide a picture of patients' function of platelet. Based on the primary result of our derivation cohort(NCT03281278), ACLF patients with high ADP inhibition rate had high 28-day mortality.This multicenter validation cohort aims to validate the predictive role of platelet mapping in ACLF prognosis, organ failure developments and short term mortality.

ELIGIBILITY:
Inclusion Criteria:

* INR≥1.5 and total bilirubin≥85μmol/L

Exclusion Criteria:

* INR≤1.5 or total bilirubin≤85μmol/L;
* those who had hepatocellular carcinoma or other types of malignancies;
* obstructive biliary diseases or other disease lead to bilirubin evaluation;
* those who had acute hemorrhage one week before admission
* those who received platelet, cryo transfusion or plasmapheresis one week before admission
* pregnancy and breastfeeding
* those who received liver transplantation or kidney transplantation;
* combine with other disease lead to organ failure including heart failure (NYHA IV),respiratory failure（PaO2<60mmHg),renal insufficiency(CKD 5) and conscious disturbance (GCS<8)
* readmission;
* death within 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACLF regardless of aetiology, International Normalized Ratio (INR)≥1.5 and total bilirubin≥85μmol/L
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-08-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28-day
  death within 28-day

SECONDARY OUTCOMES:
28-day progression | 28-day
  progressed to EASL defined ACLF
90-day mortality | 90-day
  death within 90-day

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China